CLINICAL TRIAL: NCT00998101
Title: A Phase II Trial of Carboplatin, Ixabepilone and Cetuximab in Chemotherapy Naive Advanced Non-Small Cell Lung Cancer
Brief Title: Carboplatin, Ixabepilone, and Cetuximab in Patients With Stage III or Stage IV Non-Small Cell Lung Cancer Previously Untreated With Chemotherapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was withdrawn due issuses related to the science
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0816; P30CA016086 (NIH); CDR0000656960 (Other: PDQ number)
Record Dates: First submitted 2009-10-17; First posted 2009-10-20 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cetuximab; Carboplatin; ixabepilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cetuximab — 400 mg/m2 Cycle 1 day 1 only over 120 minutes 250 mg/m2 Cycle 1 days 8,15 AND on all other cycles days 1,8,15 over 60 minutes
  Other Names: Erbitux
Drug: carboplatin — AUC=6 Day 1 of treatment over 30 minutes every 21 days
Drug: ixabepilone — 30 mg/m2 , Day 1 over 3 hours every 21 days

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin and ixabepilone, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block cancer growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry cancer-killing substances to them. Giving chemotherapy together with monoclonal antibodies may be a better way to block cancer growth.

PURPOSE: This phase II trial is studying the side effects and how well giving carboplatin and ixabepilone together with cetuximab works in treating patients with stage III or stage IV non-small cell lung cancer previously untreated with chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To estimate the disease-control rate in patients with advanced chemotherapy-naive non-small cell lung cancer after 2 courses of carboplatin, ixabepilone, and cetuximab.

Secondary

* To estimate the progression-free survival of patients treated with this regimen.
* To estimate the overall survival of patients treated with this regimen.
* To estimate the toxicity of this regimen in these patients.
* To determine the potential predictive marker of efficacy of ixabepilone and cetuximab. (exploratory)
* To investigate the prevalence of cetuximab IgE antibody, and the rate of cetuximab hypersensitivity reactions in patients without evidence of cetuximab IgE antibodies.

OUTLINE: This is a multicenter study.

Patients receive carboplatin IV over 30 minutes and ixabepilone IV over 3 hours on day 1 and cetuximab IV over 1-2 hours on days 1, 8 and 15. Treatment repeats every 21 days for up to 2-4 courses in the absence of disease progression or unacceptable toxicity. Treatment modifications may apply according to response.

Tumor tissue and blood samples are collected for further analysis.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer

  * Chemotherapy-naive
  * Stage IIIB disease not amenable to surgery with pleural effusion, pericardial effusion, or not a candidate for chemoradiotherapy
  * Stage IV disease
* Must have pathology block or unstained slides from initial or subsequent diagnosis

  * Diagnosis made via a core biopsy (not a fine-needle aspirate) required
* Measurable disease as defined by RECIST guidelines

  * For patient who received prior radiotherapy, evaluable disease must be outside of the radiation field, or have new lesions that developed within the radiation field
* Brain metastasis allowed provided it has been treated and determined to be controlled by the treating physician
* No IgE cetuximab antibody

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8.0 g/dL
* Creatinine < 2.0 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN (≤ 5 times ULN in the presence of hepatic metastasis)
* Bilirubin ≤ 1.5 times ULN
* Prior malignancy allowed provided the treating physician determines that the patient's life expectancy is best defined by diagnosis of non-small cell lung cancer (NSCLC)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No peripheral neuropathy ≥ grade 2 by NCI CTCAE v. 3.0
* No prior severe allergic reaction to any of the following:

  * Carboplatin
  * Taxane therapy
  * Monoclonal antibody
  * Hypersensitivity (NCI CTCAE grade3-4) to a drug formulated in Cremophor® EL (polyoxyethylated castor oil)
* No active or uncontrolled infection
* No significant history of uncontrolled cardiac disease including, but not limited to, any of the following:

  * Uncontrolled hypertension
  * Unstable angina
  * Myocardial infarction within the past 6 months
  * Uncontrolled congestive heart failure
  * Cardiomyopathy with decreased ejection fraction
* No underlying interstitial lung disease

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 1 week since prior and no concurrent therapeutic radiotherapy

  * Palliative radiotherapy for painful bone lesions allowed
* At least 6 months since prior adjuvant chemotherapy
* No investigational agent(s) within the past 30 days
* Not requiring concurrent treatment with any of the following:

  * Ketoconazole
  * Itraconazole
  * Ritonavir
  * Amprenavir
  * Indinavir
  * Nelfinavir
  * Delavirdine
  * Voriconazole
* No other concurrent chemotherapy or cetuximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Disease-control rate after 2 courses of carboplatin, cetuximab, and ixabepilone | 42 days
  Disease control rate will be defined as patients experiencing a complete or partial response or stable disease (radiographic response) measured by RECIST criteria.

SECONDARY OUTCOMES:
Progression-free survival | 2 years
  Radigoraphic response of measurable disease will be assessed using RECIST critera
Overall survival | 4 years
  Radigoraphic response of measurable disease will be assessed using RECIST criteria
Number of subjects experiencing adverse events | 1 year
  Adverse events will be assessed (graded) using CTCAE criteria

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Stinchcombe, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center